CLINICAL TRIAL: NCT01335217
Title: Trigeminal Nerve Stimulation for PTSD and Depression
Brief Title: Trigeminal Nerve Stimulation for Post Traumatic Stress Disorder (PTSD) and Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Ian A. Cook, M.D., Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-000894; 10-000894 (Other: UCLA Medical IRB 3)
Record Dates: First submitted 2011-04-05; First posted 2011-04-14 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Depression; Post-traumatic Stress Disorder
Keywords: Depression; Major Depressive Disorder (MDD); Trigeminal Nerve Stimulation; Post Traumatic Stress Disorder
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label TNS treatment (Other): There is only one arm in this open label treatment of MDD co-occuring with PTSD.
  Interventions: Procedure: Transcutaneous Electrical Nerve Stimulator (TENS)

INTERVENTIONS:
Procedure: Transcutaneous Electrical Nerve Stimulator (TENS) — External trigeminal nerve stimulation (TNS) as an adjunctive treatment for adults with major depressive disorder (MDD) co- occurring with posttraumatic stress disorder (PTSD) when added onto antidepressant medications

SUMMARY:
This is a 20-subject, dose finding study to examine the use of external trigeminal nerve stimulation (TNS) as an adjunctive treatment for adults with major depressive disorder (MDD) co- occurring with posttraumatic stress disorder (PTSD) when added onto antidepressant medications. Our primary objective is the examination of TNS in this patient population.

To accomplish our specific aims, the investigators will test the following specific hypotheses:

1. Subjects will show improvement in ratings of mood, PTSD, and other symptoms during the eight-week period.
2. Subjects will show improvement in ratings of life functional capacity and quality of life with TNS.
3. Subjects will report the TNS treatments to be acceptable in terms of side effects and burden of using the device.

DETAILED DESCRIPTION:
A total of 20 subjects with Major Depressive Disorder (MDD) co-occurring with Post Traumatic Stress Disorder (PTSD), ages 18 to 75 years, will be consented and join this project at UCLA.

The project will use TNS in under open-label conditions, using the same stimulation parameters as have been used in prior studies in MDD by itself and in treatment-refractory epilepsy. Subjects will be seen every two weeks during the 8 week study. At the end of the 8 weeks, the TNS systems will be returned and the adjunctive treatment will end. The co-primary endpoints are the changes in depression severity and in PTSD severity from enrollment to the week 8 visit.

ELIGIBILITY:
Inclusion Criteria

1. Outpatients with non-psychotic, unipolar Major Depressive Disorder AND Posttraumatic Stress Disorder, assessed via the MINI structured interview
2. A score of ≥ 14 on the HAM-D17 with Item 1 (depressed mood) ≥ 2
3. A score of ≥ 50 on the CAPS (Clinical-Administered PTSD Scale for DSM-IV)
4. A history of treatment failure with at least one adequate trial of an antidepressant over the previous 6 weeks, with no change in antidepressant medication or dose within the previous 6 weeks, and ongoing use of at least one antidepressant (which will continue during participation in the study)
5. Age range: 18 to 75. 6) Patients with suicidal ideation are eligible only if the thoughts of death or of life not being worth living are not accompanied by a plan or intention for self-harm.

Exclusion Criteria

1. Patient is mentally or legally incapacitated, unable to give informed consent.
2. Patients with psychosis (psychotic depression, schizophrenia, or schizoaffective diagnoses (lifetime)); bipolar disorder (lifetime); dementia (lifetime); delirium or any substance abuse disorder within the past 6 months; eating disorder within the past year; obsessive- compulsive disorder (lifetime); acute risk for suicide or self-injurious behavior. Patients with diagnostic uncertainty or ambiguity (e.g. rule-out pseudodementia of depression) will be excluded.
3. Patients with exposure to ECT or VNS within the past 6 months.
4. Past history of skull fracture; cranial surgery entering the calvarium; space occupying intracranial lesion; stroke, CVA, or TIAs; cerebral aneurysm; Parkinson's or Huntington's disease; or Multiple Sclerosis.
5. current pregnancy, breast feeding, plans to become pregnant in the 12-week treatment phase of the study, or not using a medically accepted means of contraception.
6. Other medical contraindications to any of the study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale-17 Item | Baseline, week 8
Change in PTSD Checklist score | Baseline, Week 8

SECONDARY OUTCOMES:
Change in life functional capacity and quality of life scales | baseline, week 8
  Life functional capacity and quality of life scales include: Short-form Health Survey-36 Item and Quality of Life Enjoyment and Satisfaction Questionnaire
Changes in vital signs recordings | At every visit for 8 weeks
  Autonomic function (i.e. pulse and blood pressure) are monitored for 30 mins of stimulation at baseline. Resting vital signs are recorded for each visit.
Changes in Safety Assessment Measures | At every visit for 8 weeks
  Safety Assessment measures will be administered at each visit and include: Survey of Acceptability of TNS, Systematic Assessment for Treatment Emergent Events-Systematic Inquiry (SAFTEE-SI), and Frequency, Intensity, and Burden of Side Effects Scale (FIBSER)

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Cook, M.D., Principal Investigator — Semel Institute for Neuroscience and Human Behavior
Locations (1):
- Semel Institute for Neuroscience and Human Behavior at UCLA, Los Angeles, California, United States